CLINICAL TRIAL: NCT06916390
Title: Guselkumab Intervention and Diet Evaluation for Pouchitis
Acronym: GUARDIAN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUARDIAN
Record Dates: First submitted 2025-03-21; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Pouchitis
Keywords: pouchitis; guselkumab; high fruit diet; low intake of NOVA 4 food products
MeSH Terms: conditions — Pouchitis | interventions — guselkumab; Diet

STUDY DESIGN:
Intervention Model Description: This will be a prospective, open label, parallel group, single center, randomized, (1:1) exploratory, efficacy trial at UZ Leuven.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention with guselkumab (Active Comparator): All patients will receive guselkumab 400 mg intravenous at week 0, week 4, and week 8, followed by subcutaneous guselkumab 200 mg at week 12, week 16, week 20, week 24, week 28, week 32, week 36, week 40, week 44, and week 48.
  All subjects will receive concomitant antibiotic treatment with ciprofloxacin 500mg twice daily from randomization through week 4.
  Interventions: Drug: Guselkumab
- intervention with guselkumab and diet (Active Comparator): All patients will receive guselkumab 400 mg intravenous at week 0, week 4, and week 8, followed by subcutaneous guselkumab 200 mg at week 12, week 16, week 20, week 24, week 28, week 32, week 36, week 40, week 44, and week 48.
  All subjects will receive concomitant antibiotic treatment with ciprofloxacin 500mg twice daily from randomization through week 4.
  Subjects randomized to the group with the dietary intervention will be advised to follow a low-UPF, high-fruit diet. Patients will be instructed to restrict the intake of NOVA 4 food products during the first 16 weeks of the trial, and to increase the intake of fruits (minimum 3 servings per day) during the full trial. Dietary education will be provided by certified IBD dietitians, lists of products to avoid, and week menu's will also be provided to increase dietary adherence. Dietary information will be collected with food records and food frequency questionnaires.
  Interventions: Drug: Guselkumab; Other: Diet

INTERVENTIONS:
Drug: Guselkumab — All patients will receive guselkumab 400 mg intravenous at week 0, week 4, and week 8, followed by subcutaneous guselkumab 200 mg at week 12, week 16, week 20, week 24, week 28, week 32, week 36, week 40, week 44, and week 48.
  All subjects will receive concomitant antibiotic treatment with ciprofloxacin 500mg twice daily from randomization through week 4.
  Other Names: Tremfya
Other: Diet — Subjects randomized to the group with the dietary intervention will be advised to follow a low-UPF, high-fruit diet. Patients will be instructed to restrict the intake of NOVA 4 food products during the first 16 weeks of the trial, and to increase the intake of fruits (minimum 3 servings per day) during the full trial. Dietary education will be provided by certified IBD dietitians, lists of products to avoid, and week menu's will also be provided to increase dietary adherence. Dietary information will be collected with food records and food frequency questionnaires.
  Arms: intervention with guselkumab and diet

SUMMARY:
Restorative proctocolectomy (RPC) with ileal pouch-anal anastomosis (IPAA) is considered the procedure of choice in patients with ulcerative colitis (UC) refractory to medical therapy or with neoplasia. The most common complication after IPAA is the development of pouchitis. Pouchitis is clinically characterized by variable symptoms including increased stool frequency, altered consistency, bloody stools, abdominal cramping, urgency, and incontinence. Symptomatic pouchitis longer than four weeks is considered chronic pouchitis.

The conventional treatment for acute and chronic pouchitis is antibiotics, such as metronidazole and ciprofloxacin. The disease course of antibiotic responsive pouchitis may evolve into antibiotic dependent (requiring antibiotic maintenance therapy) pouchitis and then antibiotic refractory (no response to antibiotic treatment) pouchitis. Although many patients respond to antibiotic therapy, there is also evidence that suggest that aberrant regulation of the mucosal immune system might play a part in the pathogenesis of pouchitis arising from an abnormal mucosal immune response to a dysbiosis of the pouch microbiota. If individuals fail to respond to antibiotics, anti-tumor necrosis factor (anti-TNF) agents and vedolizumab have been proposed for the treatment of chronic pouchitis.

Guselkumab, an interleukin-23 (IL-23) p19 subunit antagonist monoclonal antibody, is proven to be efficacious in patients with moderately-to-severely active UC. Efficacy of guselkumab in treating UC has been shown in multiple large clinical trials. However, patients with pouchitis were never the targeted population and were even often excluded from the trials.

Pouchitis becomes a chronic problem with a huge impact in the quality of life of these patients. The incidence of pouchitis has been rising in the last decades. This increase might be explained by a change in dietary habits of this population.

This open label single center trial at UZ Leuven aims to evaluate the efficacy and safety of guselkumab in the treatment of chronic antibiotic refractory pouchitis during a 48-week treatment period, with or without a dietary intervention. Twenty subjects with a proctocolectomy and IPAA for UC who have developed chronic or relapsing pouchitis will be enrolled.

DETAILED DESCRIPTION:
Restorative proctocolectomy (RPC) with ileal pouch-anal anastomosis (IPAA) is considered the procedure of choice in patients with ulcerative colitis (UC) refractory to medical therapy or with neoplasia. The most common complication after IPAA is the development of pouchitis. Pouchitis is clinically characterized by variable symptoms including increased stool frequency, altered consistency, bloody stools, abdominal cramping, urgency, and incontinence. Between 50% and 80% of those with an IPAA will experience pouchitis symptoms at any given moment with 10% of patients developing a chronic antibiotic refractory pouchitis. Symptomatic pouchitis for less than four weeks is considered acute pouchitis, while symptomatic pouchitis longer than four weeks is considered chronic pouchitis. Additionally, relapsing pouchitis can also occur when there are three or more episodes per year.

The conventional treatment for acute and chronic pouchitis is antibiotics, such as metronidazole and ciprofloxacin. The clinical response of pouchitis to treatment with antibiotics such as metronidazole or ciprofloxacin, suggests that fecal stasis, Clostridium difficile infection, bacterial overgrowth or dysbiosis (qualitative or quantitative alterations in the bacterial communitiy) may be triggers. The disease course of antibiotic responsive pouchitis may evolve into antibiotic dependent (requiring antibiotic maintenance therapy) pouchitis and then antibiotic refractory (no response to antibiotic treatment) pouchitis. Although many patients respond to antibiotic therapy, there is also evidence that suggest that aberrant regulation of the mucosal immune system might play a part in the pathogenesis of pouchitis arising from an abnormal mucosal immune response to a dysbiosis of the pouch microbiota. If individuals fail to respond to antibiotics, anti-tumor necrosis factor (anti-TNF) agents and vedolizumab have been proposed for the treatment of chronic pouchitis. Recently, vedolizumab has been shown to be efficacious in treating chronic pouchitis with remission rates of 31% at week 14. Nevertheless, the treatment of chronic pouchitis remains an unmet need for patients with inflammatory bowel diseases (IBD).

Guselkumab, an interleukin-23 (IL-23) p19 subunit antagonist monoclonal antibody, is proven to be efficacious in patients with moderately-to-severely active UC. In the phase II GALAXI 1 trial (309 patients with UC, 2020), intravenous treatment with 200 mg, 600 mg or 1,200 mg guselkumab at weeks 0, 4 and 8 showed significantly greater reductions from baseline CDAI, outcomes of clinical response, clinical remission, Patient-Reported Outcome-2 (PRO-2) remission, clinical biomarker response and endoscopic response at week 12 compared with intravenous placebo. The QUASAR study (313 patients with UC, 2022), a Phase 2b/3 randomized, double-blind, placebo-controlled trial, demonstrated superiority of guselkumab to placebo for clinical response during induction at week 12 in patients with UC. Guselkumab also met key secondary endpoints of clinical remission, symptomatic remission, endoscopic improvement, and histo-endoscopic mucosal improvement. The efficacy and safety of guselkumab in patients with UC were further studied in the exploratory Phase 2a VEGA trial (214 patients with UC, 2023) evaluating combination treatment of guselkumab and golimumab during induction. Combination therapy was significantly more effective than either drug alone for clinical remission and endoscopic improvement. A meta-analysis (36 studies with 14270 patients with UC, 2024) comparing the relative efficacy of biologics and small molecules, proved Guselkumab to rank high in achieving clinical remission, endoscopic improvement and remission, and histological remission in patients with moderate to severe UC. Efficacy of guselkumab in treating UC has been shown in multiple large clinical trials. However, patients with pouchitis were never the targeted population and were even often excluded from the trials.

Pouchitis becomes a chronic problem with a huge impact in the quality of life of these patients. The incidence of pouchitis has been rising in the last decades. This increase might be explained by a change in dietary habits of this population. Interestingly, lower fruit consumption has been associated with higher risk of pouchitis. Moreover, food colorants have been associated with colitis in mice with higher IL-23 expression.

This open label single center trial at UZ Leuven aims to evaluate the efficacy and safety of guselkumab in the treatment of chronic antibiotic refractory pouchitis during a 48-week treatment period, with or without a dietary intervention. Twenty subjects with a proctocolectomy and IPAA for UC who have developed chronic or relapsing pouchitis will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. At least 18 years of age at the time of signing the Informed Consent Form (ICF)
3. Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.
4. Participant with a proctocolectomy and IPAA for UC who heveloped chronic or relapsing pouchitis, defined as mPDAI score ≥5 and a minimum endoscopic subscore of 2 (outside the staple or suture line) with either:

   1. ≥2 recurrent episodes within 1 year prior to the screening visit, each treated with ≥2 weeks of antibiotic or other prescription therapy, or
   2. patients treated with maintenance antibiotic therapy taken continuously for four consecutive weeks before the screening visit and who are refractory to this antibiotic therapy, or
   3. previously failure of another biologic therapy to treat chronic pouchitis.
5. The subject agrees to take ciprofloxacin (500 mg twice daily) on Day 1 and through Week 4, regardless of the previous treatment and to stop any previous antibiotic therapy on Day 1 of the study. For patients who did previously not tolerate quinolone therapy, an alternative antibiotic therapy between Day 1 and Week 4 with metronidazole (500 mg three times a day) will be allowed. (Additional courses of antibiotics will be allowed, as needed, for flares after Week 16.)

All participants that are considered for Trial participation, per the above criteria will be documented via applicable log forms in Investigator Site File (including Screen Failures).

Exclusion Criteria:

1. Crohn's disease (CD), CD-related complications of the pouch (pouch fistula, pouch strictures, ulcerations in the pre-pouch ileum without pouchitis), irritable pouch syndrome (IPS), isolated or predominant cuffitis, infectious pouchitis, diverting ostomy or mechanical complications of the pouch
2. Previous treatment with an anti-IL12/23 or an anti-IL23 antibody
3. Any investigational or approved biologic agent within 30 days of screening
4. Nonbiologic investigational therapy or JAK inhibitors within 30 days prior to screening
5. Active or untreated latent tuberculosis (TB). In case of a newly identified positive diagnostic TB test result (defined as a positive tuberculin skin test) , active TB has to be ruled out and appropriate treatment for latent TB has to be initiated for a minimum of 4 weeks prior to the first administration of study medication.
6. Chronic hepatitis B virus (HBV)* infection, chronic hepatitis C virus (HCV)** infection, a known history of human immunodeficiency virus (HIV) infection (or is found to be seropositive at screening) or subject is immunodeficient (e.g., due to organtransplantation, history of common variable immunodeficiency, etc). * Subjects who are positive for hepatitis B virus surface antigen (HBsAg) will be excluded. For subjects who are negative for HBsAg but are positive for either surface antibodiesand/or core antibodies, HBV DNA polymerase chain reaction will be performed and if anytest result meets or exceeds detection sensitivity, the subject will be excluded.** If subject is HCV antibody positive, then a viral load test will be performed. If the viralload test is positive then the subject will be excluded.
7. Active severe infection (eg sepsis, cytomegalovirus, listeriosis or C. difficile)
8. The subject has allergies to and/or contraindications for ciprofloxacin and metronidazole
9. Participant has a history of malignancy or current malignancy, except for the following: adequately treated non-metastatic basal cell skin cancer, squamous cell skin cancer and cervical carcinoma in situ. Subjects with a remote history of malignancy (e.g., >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy.
10. Any disorder or laboratory abnormalities which in the Investigator's opinion might jeopardise the participant's safety or compliance with the protocol.
11. Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial (see list in 5.3).
12. Female who is pregnant, breast-feeding or intends to become pregnant before, during, or within 15 weeks after the last dose of study drug; or intending to donate ova during such time period or is of child-bearing potential and not using an adequate, highly effective contraceptive or males who want to make their partner pregnant or intends to donate sperm during the course of this study or for 18 weeks after the last dose of study drug
13. Participation in another interventional Trial with an investigational medicinal product (IMP) or device.

Participants who meet one or more of the above exclusion criteria must not proceed to be enrolled/randomized in the Trial and will be identified via applicable log forms in Investigator Site File.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
percentage of subjects achieving clinical remission after 16 weeks of treatment with guselkumab with/without diet | 16 weeks
  the percentage of subjects with chronic or recurrent pouchitis achieving clinical remission (mPDAI score <5 and a reduction of overall score by ≥2 points from Baseline) after 16 weeks of treatment with guselkumab compared to 16 weeks of guselkumab and a dietary intervention.

SECONDARY OUTCOMES:
percentage of subjects achieving clinical remission after 48 weeks | 48 weeks
  The percentage of subjects achieving clinical remission (mPDAI score <5 and a reduction of overall score by ≥2 points from Baseline) after 48 weeks in both groups
percentage of subjects achieving antibiotic free clinical remission by week 16 and 48 | week 16 and week 48
  The percentage of subjects achieving antibiotic free clinical remission by week 16 and 48
percentage of subjects achieving partial response after 16 and 48 weeks | week 16 and week 48
  The percentage of subjects achieving partial response (reduction of mPDAI score by ≥2 points from Baseline) after 16 and 48 weeks in both groups
Time to clinically relevant remission | 48 weeks
  Time to clinically relevant remission in both groups
Change in mPDAI endoscopic subscore at Week 16 and 48 | baseline, week 16 and week 48
  Change in mPDAI endoscopic subscore at Week 16 and 48 compared to Baseline in both groups
Change in mPDAI histologic subscore at Week 16 and 48 | baseline, week 16 and week 48
  Change in mPDAI histologic subscore at Week 16 and 48 compared to Baseline in both groups
Change in total mPDAI score at Week 16 and 48 | baseline, week 16 and week 48
  Change in total mPDAI score at Week 16 and 48 compared to Baseline in both groups
percentage of subjects achieving a flare after initial response | 48 weeks
  The percentage of subjects achieving a (endoscopic proven) flare after initial response in both groups
Microbiota Metagenomic profiling at Week 8, 16, 24, 32, 40 and 48 | baseline, week 8, 16, 24, 32, 40 and week 48
  Microbiota Metagenomic profiling (changes in intestinal microbiota) at Week 8, 16, 24, 32, 40 and 48 compared to Baseline in both groups
Changes in IL-23p19 expression in the tissue at Week 16 and 48 | baseline, week 16 and week 48
  Changes in IL-23p19 expression in the tissue at Week 16 and 48 compared to Baseline in both groups
Statistical association between IL-23p19 expression and response to therapy | 48 weeks
  Statistical association between IL-23p19 expression and response to therapy in both groups
Food record and food frequency questionnaire | 48 weeks
  Food record and food frequency questionnaire in the group with the dietary intervention
adverse event assessment of interventions | 48 weeks
  adverse event assessment of the interventions
questionnaire about diet tolerability | 48 weeks
  questionnaire about tolerability of the prescribed diet in the group with the dietary intervention

OTHER OUTCOMES:
Time to relapse of pouchitis symptoms and number of relapses | 48 weeks
  Time to relapse of pouchitis symptoms and number of relapses in both groups
Change in CRP at Week 8, 16, 24, 32, 40 and 48 | baseline, week 8, 16, 24, 32, 40 and week 48
  Change in CRP at Week 8, 16, 24, 32, 40 and 48 compared to Baseline in both groups
Change in faecal calprotectin at Week 8, 16, 24, 32 and 48 | baseline, week 8, 16, 24, 32, 40 and week 48
  Change in faecal calprotectin at Week 8, 16, 24, 32 and 48 compared to Baseline in both groups
Evolution of guselkumab serum levels | baseline, week 8, 16, 24, 32, 40 and week 48
  Evolution of guselkumab serum levels between Baseline and Week 8, 16, 24, 32, 40 and 48 in both groups
Evolution of anti-guselkumab antibodies | baseline, week 8, 16, 24, 32, 40 and week 48
  Evolution of anti-guselkumab antibodies between Baseline and Week 8, 16, 24, 32, 40 and 48 in both groups
Statistical correlation of guselkumab serum levels and anti-guselkumab antibodies with clinical, endoscopic and histological outcomes | baseline, week 8, 16, 24, 32, 40 and week 48
  Statistical correlation of guselkumab serum levels and anti-guselkumab antibodies with clinical, endoscopic and histological outcomes between Baseline and Week 8, 16, 24, 32, 40 and 48 in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- university hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No